CLINICAL TRIAL: NCT00716378
Title: Teenage Passenger Influences on the Simulated Driving Performance of Teenage Drivers
Brief Title: Teenage Passenger Influences on Driving Performance of Teenage Drivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 999908183; 08-CH-N183
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-11-15

CONDITIONS: Motor Vehicle Crash Injuries
Keywords: Simulated Driving; Risky Driving Behavior; Social Influences

INTERVENTIONS:
Behavioral: Teen Passenger Presence

SUMMARY:
This study, conducted at the University of Massachusetts at Amherst, will examine how male teenage driving performance varies in the presence or absence of male teenage passengers. It will explore what information teen drivers and their passengers use when making decisions that affect their performance on the road.

Male drivers under 18 years of age who have a Junior Operator's or Full License and have driven at least once in the month before enrolling in the study may be eligible to participate.

In a university laboratory, participants sit in a 1995 Saturn sedan and operate the controls of the car just as they would those of any other car, during simulated drives in urban, suburban and rural areas. They are fitted with a head-mounted eye tracker that records their point of gaze in real time. On one drive, the subject drives alone; on another, a male passenger rides along. After the drives, the subject fills out some questionnaires.

DETAILED DESCRIPTION:
The purpose of this research is to examine how male teenage driving performance varies in the presence or absence of high versus low risk accepting male teenage passengers. Driving performance includes attention and risk measures including eye glance behaviors, speed management, following distance, closing speed and gap acceptance. To what extent does driving performance vary as a product of the male teen passenger risk- acceptance compared with no passenger present?

ELIGIBILITY:
* INCLUSION CRITERIA:

Only male driver and passengers

Under the age of 18

Having a provisional or full license (i.e. allowing driving without supervision)

Having driven in the past 3 months

Having normal or corrected-to-normal vision (i.e. contact lenses or eye glasses are accepted)

EXCLUSION CRITERIA:

Females

Motion sickness

Ages: 16 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2008-07-11; Primary Completion 2010-11-15 (Actual); Study Completion 2010-11-15 (Actual)

PRIMARY OUTCOMES:
Risky Driving Behavior

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), 9000 Rockville, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chen LH, Baker SP, Braver ER, Li G. Carrying passengers as a risk factor for crashes fatal to 16- and 17-year-old drivers. JAMA. 2000 Mar 22-29;283(12):1578-82. doi: 10.1001/jama.283.12.1578. PMID 10735394
- [Background] Dielman TE, Campanelli PC, Shope JT, Butchart AT. Susceptibility to peer pressure, self-esteem, and health locus of control as correlates of adolescent substance abuse. Health Educ Q. 1987 Summer;14(2):207-21. doi: 10.1177/109019818701400207. PMID 3597110
- [Background] Fisher DL, Pollatsek AP, Pradhan A. Can novice drivers be trained to scan for information that will reduce their likelihood of a crash? Inj Prev. 2006 Jun;12 Suppl 1(Suppl 1):i25-9. doi: 10.1136/ip.2006.012021. PMID 16788108